CLINICAL TRIAL: NCT03474770
Title: Evaluation of Safety and Efficacy of BIS-001-ER for the Treatment of Adult Focal Impaired Awareness Seizures
Brief Title: BIS-001-ER for the Treatment of Adult Focal Impaired Awareness Seizures
Acronym: FIAS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNI-02-1b
Record Dates: First submitted 2018-03-12; First posted 2018-03-23 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Focal Impaired Awareness Seizures
MeSH Terms: conditions — Seizures | interventions — huperzine A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIS-001ER (Experimental): Dose administration for each participant will begin at 0.25mg b.i.d. escalating sequentially every 4 days to a maximum tolerated dose or target dose of 1.75mg b.i.d. Upon reaching the target dose or maximum tolerated dose, participants will maintain that dose for the balance of the 1 month out-patient titration period, after which they will begin a 96-hour in-patient video EEG monitoring treatment period.
  Interventions: Drug: BIS-001ER

INTERVENTIONS:
Drug: BIS-001ER — BIS-001 ER is an extended release formulation of the nutritional supplement Huperzine A.
  Other Names: Huperzine A ER

SUMMARY:
The purpose of this study is to examine safety signals and demonstrate seizure reduction in adults with FIAS treated with BIS-001ER as an add-on therapy in an in-patient and out-patient study design.

ELIGIBILITY:
Inclusion Criteria:

* Speak English with sufficient proficiency to read and comprehend the Informed Consent document, and to communicate with study staff.
* Be able to consent to participate by signing the Informed Consent document after a full explanation of the nature and purpose of this study.
* Have signed the Informed Consent before any study-specific procedures are performed.
* Be males or females between 18 - 65 years of age.
* Have a diagnosis of FIAS type epilepsy with or without additional focal aware or non-aware seizures with generalization.
* Have a current minimum average of 5 countable seizures / week to enroll in study.
* Have at least 5 focal impaired awareness seizures during the 96-hour baseline VEM period.
* Be receiving stable doses (for at least 4 weeks) of one to four currently marketed anti-epileptic drugs (AEDs), with or without vagus nerve stimulation (in which case the patient should be on the same stimulation parameters for at least 4 weeks).
* Have a negative urinary pregnancy test upon admission to the site on Day 1.
* Be in good general health in the judgment of the Principal Investigator based upon medical history, physical examination, standard 12-lead ECG, and clinical laboratory evaluations obtained within the two weeks prior to enrollment.
* Be able to comply with all study-specified procedures.
* Weight between 40 and 120 kg.

Exclusion Criteria:

* Has taken Huperzine A within the past year.
* Is planning to become pregnant or impregnate spouse, not using an acceptable method of birth control (defined as use of double-barrier birth control methods, use of oral contraceptives, or surgical sterilization), pregnant or nursing.
* Have non-epileptic events that could be confused by the patient and/or study staff as epileptic seizures.
* Has seizures that are difficult to count; for example, seizure clusters defined as multiple seizures with at least one seizure within 30 minutes of the previous seizure.
* Have less than the 5 minimum accepted seizures required during baseline evaluation period screen.
* Have a history of only seizure clusters, for example, seizure clusters defined as multiple seizures with at least one seizure within 30 minutes of the previous seizure.
* Has attempted suicide within the past 2 years.
* Has a history of status epilepticus in the 6 months previous to enrollment.
* Has a pre-existing medical condition (including an existing progressive or degenerative neurological disorder including brain tumor, active encephalitis, active meningitis or abscess) or takes medications that, in the Principal Investigator's opinion, could interfere with the participant's suitability for participation in the study.
* Has a history or evidence of significant psychiatric disturbance or illness, including alcohol or drug abuse within the past 2 years, or symptoms of psychosis (hallucinations, delusions) in the last 5 years.
* Has had any clinical laboratory abnormalities within the past two months, prior to screening, considered of clinical significance by the Principal Investigator.
* Is on concomitant therapy with non-AEDs that are cholinergic.
* Has participated in any clinical investigational drug or device study within four weeks prior to study entry.
* Inability to complete seizure diary.
* Is currently taking or has taken Epigallocatechin gallate (EGCG) within the past 14 days, or consume foods or drinks containing EGCG; including green, white, oolong teas and certain black teas, or food containing >100grams of carob powder within the past 14 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Effect of BIS-001ER on Seizure Count | 6 Weeks
  Reduction in average daily seizure count between baseline (pre-treatment) and evaluation (on treatment) video EEG monitoring periods.

SECONDARY OUTCOMES:
Effect of BIS-001ER on Percent Reduction in Daily Seizure Count | 6 Weeks
  Percent reduction in average daily seizure count from the baseline VEM period compared to the evaluation video EEG monitoring period (on treatment).
Effect of BIS-001ER on Seizure Count vs Titration Period (Diary) | 6 Weeks
  Percent reduction in average number of seizures from the baseline period. (screening/retrospective diary) compared to the last week of the titration treatment period.
Percent of Treatment Responders | 6 Weeks
  Percent of participants considered treatment responders defined as those with a ≥25%, ≥50%, ≥75% reduction in seizures from the baseline VEM period compared to the VEM treatment evaluation period.
Effect of BIS-001ER on Seizure Count During Extension Phase | 12 Months
  Percent reduction of average number of seizures vs. baseline/retrospective diary at 1, 3, 6, 12 months during the extension period.
Complete Seizure Protection | 6 Weeks
  Proportion of subjects with 100% seizure reduction.
Need for Rescue Medication | 6 Weeks
  Proportion of subjects requiring rescue medication at different dosages.

CONTACTS AND LOCATIONS:
Overall Officials: Azmi Nasser, PhD, Study Chair — Supernus Pharmaceuticals, Inc.
Locations (2):
- Australia (2):
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria